CLINICAL TRIAL: NCT01177969
Title: CBT for Anxiety Disorders in Autism: Adapting Treatment for Adolescents
Brief Title: Cognitive Behavioral Therapy (CBT) for Anxiety Disorders in Autism: Adapting Treatment for Adolescents
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of California, Los Angeles (Other); University of Miami (Other)
Responsible Party: Principal Investigator, Eric Storch, Professor, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R34HD065274-01 (NIH); 1R34HD065274-01 (NIH)
Record Dates: First submitted 2010-08-05; First posted 2010-08-09 (Estimated); Results first posted 2014-07-01 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Anxiety Disorders in Youth With Autism, Asperger's Syndrome, and Pervasive Developmental Disorder Not Otherwise Specified
Keywords: Autism; Anxiety; Asperger's Syndrome; Cognitive-behavioral therapy; Treatment; Obsessive-compulsive disorder; Fears
MeSH Terms: conditions — Asperger Syndrome; Autistic Disorder; Anxiety Disorders; Obsessive-Compulsive Disorder | interventions — Cognitive Behavioral Therapy; Implosive Therapy; Waiting Lists

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive-Behavioral Therapy (Experimental): The form of treatment will involve 16 weekly meetings of about 90 minutes each. Sessions involve both the child and parent and involve teaching youth how to cope with their anxiety through a variety of behavioral techniques.
  Interventions: Behavioral: Cognitive-Behavioral Therapy
- Wait-list (Placebo Comparator): A wait-list essentially involves not receiving treatment for a specified period of time (in this case 16 weeks). No active treatment is provided; rather, the family 'waits'.
  Interventions: Behavioral: Wait-list

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Therapy — The form of treatment will involve 16 weekly meetings of about 90 minutes each. Sessions involve both the child and parent and involve teaching youth how to cope with their anxiety through a variety of behavioral techniques.
  Other Names: CBT; Exposure therapy
  Arms: Cognitive-Behavioral Therapy
Behavioral: Wait-list — A wait-list essentially involves not receiving treatment for a specified period of time (in this case 16 weeks). No active treatment is provided; rather, the family 'waits'.
  Other Names: Placebo
  Arms: Wait-list

SUMMARY:
Comorbid anxiety disorders affect as many as 80% of youth with autism spectrum disorders, causing substantial distress and impairment over and above the autism spectrum diagnosis alone. Cognitive behavioral therapy (CBT) is the gold standard treatment among typically developing youth with an anxiety disorder and when adapted, shows promise in children with ASD and comorbid anxiety. However, there is currently no psychotherapy protocol tailored to meet the unique needs of young adolescents with Autism spectrum disorders (ASD) and comorbid anxiety. Given this, the present study seeks to develop and test a new CBT therapy in adolescents with autism and comorbid anxiety.

DETAILED DESCRIPTION:
Autism spectrum disorders (ASD) affect approximately 1 out of 150 children and adolescents in the United States, making them one of the most common neurobiological conditions. Comorbid anxiety disorders affect as many as 80% of youth with ASD, causing substantial distress and impairment over and above that caused by an ASD diagnosis alone. While cognitive-behavioral therapy (CBT) has been established as the gold standard treatment for anxiety disorders among typically developing youth, a protocol does not exist for early adolescents with ASD and comorbid anxiety disorders. Accordingly, we are proposing to develop a CBT protocol for anxiety and comorbid ASD in early adolescence.

Initial protocol development efforts will focus on adapting relevant treatment elements from an effective CBT program for younger children with ASD and comorbid anxiety to the characteristics and clinical needs of early adolescents. Thereafter, protocol and measure development will be refined during Phases I and II of this study through our experiences treating a total of 20 young adolescents (ages 11-14 years - 10 will be treated at USF; 10 at University of California, Los Angeles (UCLA)) with ASD and comorbid anxiety disorder(s). The CBT protocol will then be examined in a trial comparing CBT to a waitlist condition (N = 32 total; 16 at each study site).

The two recruitment sites for this study are the University of California, Los Angeles and the University of South Florida. The University of Miami will assist with quality assurance checks. Considering the rising number of youth diagnosed with ASD, and the lack of tested treatment options for those young adolescents with comorbid anxiety, our proposed work toward an efficacious CBT protocol will provide a timely contribution to public health efforts.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient adolescents with ASD (see below) between the ages 11-14 years.
* Meets criteria for a diagnosis of autism, Asperger syndrome (AS), or Pervasive Developmental Disorder Not Otherwise Specified .
* Meets criteria for a diagnosis of one of the following anxiety disorders: separation anxiety disorder (SAD), generalized anxiety disorder (GAD), social phobia, or obsessive compulsive disorder (OCD).
* Child has a Full Scale and Verbal Comprehension IQ≥85.

Exclusion Criteria:

* Receiving concurrent psychotherapy, social skills training, or behavioral interventions (e.g., applied behavior analysis). Families will have the option of discontinuing such services to enroll in the study.
* Has started an antidepressant within 12 weeks before study enrollment or an antipsychotic 6 weeks before study enrollment.
* Has changed established psychotropic medications (e.g., antidepressants, anxioloytics) within 8 weeks before study enrollment (6 weeks for antipsychotic).
* Is currently suicidal or has been actively suicidal in the last 6 months.
* Has been diagnosed with bipolar, schizophrenia or schizoaffective disorders; or Substance abuse in past 6 months.
* Presence of a significant and/or unstable medical illness which might lead to hospitalization during the study.

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2009-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Storch, PhD, Principal Investigator — University of South Florida
Locations (2):
- United States (2):
  - Univeristy of California at Los Angeles, Los Angeles, California
  - University of South Florida, St. Petersburg, Florida

REFERENCES:
- [Derived] Elliott SJ, Marshall D, Morley K, Uphoff E, Kumar M, Meader N. Behavioural and cognitive behavioural therapy for obsessive compulsive disorder (OCD) in individuals with autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2021 Sep 3;9(9):CD013173. doi: 10.1002/14651858.CD013173.pub2. PMID 34693989
- [Derived] Wood JJ, Ehrenreich-May J, Alessandri M, Fujii C, Renno P, Laugeson E, Piacentini JC, De Nadai AS, Arnold E, Lewin AB, Murphy TK, Storch EA. Cognitive behavioral therapy for early adolescents with autism spectrum disorders and clinical anxiety: a randomized, controlled trial. Behav Ther. 2015 Jan;46(1):7-19. doi: 10.1016/j.beth.2014.01.002. Epub 2014 Jan 22. PMID 25526831
- See also: Related Info — http://hscweb3.hsc.usf.edu/health/now/?p=8518

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cognitive-Behavioral Therapy | Wait-list
Started | 19 | 14
Completed | 16 | 11
Not Completed | 3 | 3
Not completed — Protocol Violation | 2 | 1
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive-Behavioral Therapy | Wait-list | Total
Number analyzed (Participants) | 19 | 14 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.4 (1.3) | 12.2 (.98) | 12.3 (1.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 13 | 10 | 23
Region of Enrollment [Number; unit: participants]
  United States | 19 | 14 | 33

OUTCOME MEASURES:

1. Primary Outcome: Pediatric Anxiety Rating Scale.
Description: The Pediatric Anxiety Rating Scale is a clinician-rated scale assessing anxiety symptoms and the associated severity and impairment in children over the past week. The scale includes 5 items which are summed to form a total score, which represents anxiety severity. The scale score ranges from 0 to 25 with higher scores indicating more severe anxiety symptoms.
Time Frame: Post-treatment, which is an average of 16 weeks after Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive-Behavioral Therapy | Wait-list
Number analyzed (Participants) | 19 | 14
units on a scale | 11.62 (3.26) | 14.04 (2.64)
Statistical Analysis 1: Comparison: Cognitive-Behavioral Therapy vs Wait-list; Test type: Superiority or Other; p = .04, ANCOVA — This analysis applies to the post-treatment assessment (16 weeks after baseline)

2. Secondary Outcome: Anxiety Disorders Interview Schedule: Child and Parent Versions
Description: The Anxiety Disorders Interview Schedule: Child and Parent Versions are clinician-rated scales assessing anxiety symptoms and the associated severity and impairment in children over the past month. The clinician interviewer interviews the child and parent separately about the nature and severity of the child's anxiety. If a child meets criteria for an anxiety disorder, a single item is rated by the interviewer, which represents anxiety severity. The scale score for this single item ranges from 0 to 8 with higher scores indicating more severe anxiety symptoms.
Time Frame: Post-treatment, which was an average of 16 weeks after Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive-Behavioral Therapy | Wait-list
Number analyzed (Participants) | 19 | 14
units on a scale | 3.28 (2.1) | 4.04 (1.88)
Statistical Analysis 1: Comparison: Cognitive-Behavioral Therapy vs Wait-list; Test type: Superiority or Other; p = .25, ANCOVA — This analysis applies to the post-treatment assessment (16 weeks after baseline)

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: Queries by study staff at study visits.
Arm/Group | Cognitive-Behavioral Therapy | Wait-list
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/14
Other Adverse Events (participants affected / at risk) | 0/19 | 0/14

LIMITATIONS AND CAVEATS:
Modest sample size Lack of objective measures of anxiety that go beyond diagnostic interview or checklist measures

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No